CLINICAL TRIAL: NCT06914908
Title: A Single-arm Extension Study to Investigate the Long-term Safety, Tolerability, and Efficacy of Lunsekimig in Adult Participants With Inadequately Controlled Chronic Rhinosinusitis With Nasal Polyps (CRSwNP) Who Completed a Previous Lunsekimig CRSwNP Clinical Study
Brief Title: Long-term Safety and Efficacy Evaluation of Lunsekimig in Adult Participants With Chronic Rhinosinusitis With Nasal Polyps (CRSwNP) Who Completed a Previous Lunsekimig CRSwNP Study
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LTS18300; 2024-515912-27 (Registry Identifier: CTIS)
Record Dates: First submitted 2025-04-04; First posted 2025-04-07 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Chronic Rhinosinusitis With Nasal Polyps

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Lunsekimig (Experimental): Participant will receive lunsekimig subcutaneous (SC) every 4 weeks and intranasal mometasone furoate nasal spray (MFNS) daily for 52 weeks.
  Interventions: Drug: lunsekimig; Drug: Mometasone furoate nasal spray (MFNS)

INTERVENTIONS:
Drug: lunsekimig — Pharmaceutical form: solution for injection Route of administration: subcutaneous
  Other Names: SAR443765
Drug: Mometasone furoate nasal spray (MFNS) — Pharmaceutical form: Intranasal spray Route of administration: intranasal

SUMMARY:
This is a single-arm extension study to investigate the long-term safety, tolerability, and efficacy of lunsekimig in adult participants with inadequately controlled CRSwNP who have completed a previous lunsekimig CRSwNP clinical study (also referred to as the parent study ACT18207).

The study duration will be up to approximately 56 weeks per participant, 52 weeks of treatment period, and 4 weeks of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Participants who have completed the treatment period and the follow up period in CRSwNP lunsekimig parent study, including EOS visit, as per protocol.
* Participants receiving therapy with intranasal mometasone furoate nasal spray (MFNS).
* Participants who are able and willing to participate in this extension study, and to comply with requested study visits and procedures.

Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply:

* Prior hypersensitivity reaction to lunsekimig or to any of the excipients used in the presentation or in preparation for administration of lunsekimig, or other allergy that, in the opinion of the Investigator, contraindicates participation in the study.
* Concurrent participation in any clinical study other than the parent study, including non-interventional studies.
* Participants who, during their participation in the parent study, developed an adverse event (AE) or a serious adverse event (SAE) deemed related to lunsekimig, which in the opinion of the Investigator could indicate that continued treatment with lunsekimig may present an unreasonable risk for the participant.

NOTE: The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2025-05-12 (Actual); Primary Completion 2031-01-29 (Estimated); Study Completion 2031-01-29 (Estimated)

PRIMARY OUTCOMES:
Incidence of participants with treatment-emergent adverse events (TEAEs) including | From baseline to end of study (approximately 56 weeks)

SECONDARY OUTCOMES:
Change in SNOT-22 total score | From the parent study baseline to Week 52
  The SNOT-22 is a 22-item health-related outcomes assessment. The 22-question SNOT-22 is scored as 0 (no problem) to 5 (problem as bad as it can be) with a total range from 0 to 110 (higher scores indicate poorer outcomes).
Change in rhinosinusitis visual analog scale (VAS) | From the parent study baseline to Week 52
  The VAS for rhinosinusitis is used to evaluate the total severity. The participant is asked to indicate along a 10 centimeter straight horizontal line (VAS) the answer to the question: "How troublesome are your symptoms of your rhinosinusitis". The VAS ranks from 0 (Not troublesome) to 10 (Worst thinkable troublesome) and is measured in centimeters
Change in University of Pennsylvania Smell Identification Test (UPSIT) score | From the parent study baseline to Week 52
  The UPSIT test is a rapid and easy-to-administer method to quantitatively assess human olfactory function. The test consists of four booklets, each containing 10 odorants with one odorant per page. Above each odorant strip is a multiple-choice question with four alternative words to describe the odor. Score depends on the amount of answers out of 40 possible correct answers.
Serum lunsekimig concentrations | From baseline to end of study (approximately 56 weeks)
Anti-drug antibodies (ADA) against lunsekimig | From baseline to end of study (approximately 56 weeks)

CONTACTS AND LOCATIONS:
Locations (17):
- United States (7):
  - Modena Allergy + Asthma- Site Number : 8400005, La Jolla, California
  - Treasure Valley Medical Research- Site Number : 8400002, Boise, Idaho
  - Essential Medical Research- Site Number : 8400020, Tulsa, Oklahoma
  - McGovern Medical School - UT Physicians Dermatology - Bellaire Station- Site Number : 8400017, Bellaire, Texas
  - Pharmaceutical Research & Consulting- Site Number : 8400004, Dallas, Texas
  - ENT Associates of Texas - McKinne- Site Number : 8400014, McKinney, Texas
  - Alamo ENT Associates- Site Number : 8400001, San Antonio, Texas
- Argentina (3):
  - Investigational Site Number : 0320002, Rosario, Santa Fe Province
  - Investigational Site Number : 0320001, Buenos Aires
  - Investigational Site Number : 0320003, Mendoza
- Investigational Site Number : 0560002, Ghent, Belgium
- Investigational Site Number : 1000001, Sofia, Bulgaria
- Poland (4):
  - Investigational Site Number : 6160004, Poznan, Greater Poland Voivodeship
  - Investigational Site Number : 6160002, Krakow, Lesser Poland Voivodeship
  - Investigational Site Number : 6160007, Wroclaw, Lower Silesian Voivodeship
  - Investigational Site Number : 6160003, Katowice, Silesian Voivodeship
- Investigational Site Number : 8260001, Newcastle upon Tyne, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: LTS18300 Plain Language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=26670&tenant=MT_SNY_9011